CLINICAL TRIAL: NCT00323531
Title: Thoracoscopy Versus Fibrinolysis in Children With Empyema
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Shawn St. Peter, Children's Mercy Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06 01-019
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Empyema
Keywords: thoracoscopy; fibrinolysis; empyema; children
MeSH Terms: conditions — Empyema | interventions — Chest Tubes; Fibrinolysis; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Video assisted thoracoscopic decortication
  Interventions: Procedure: VATS decortication
- 2 (Experimental): Fibrinolysis through the chest tube
  Interventions: Procedure: Chest tube with tPA infusion for 3 days

INTERVENTIONS:
Procedure: Chest tube with tPA infusion for 3 days — fibrinolysis through the chest tube
  Other Names: Fibrinolysis; tPA
  Arms: 2
Procedure: VATS decortication — thoracoscopic decortication
  Other Names: VATS; pleural debridement
  Arms: 1

SUMMARY:
The null hypothesis is that patients receiving either thoracoscopy or fibrinolysis for empyema recover in the same amount of time. Therefore, we will test this by randomizing the next 40 patients who consent to the study to one treatment or the other.

DETAILED DESCRIPTION:
This will be a single institution, prospective, randomized clinical trial involving patients who are found to have at least a single septation within a pleural effusion as diagnosed by ultrasound or computed tomography. Additionally, patients with a pleural effusion wherein a pleural tap reveals pus as defined by many (> 10,000/mm3 ) white blood cells or positive cultures will be considered. This is intended to be a definitive study.

Power calculations based on the known 4.8 post intervention hospital days after VATS and the estimated 7 post intervention days after fibrinolysis with α = 0.05 and power of 0.8 show the need for 18 patients in each arm. We will intend to recruit 40. This sample size was constructed in consultation with Dr. Steve Simon, and the range of hospital stay in our retrospective experience was utilized. Therefore, this number should represent an adequate power in spite of the known varied level of illness.

One group will undergo thoracoscopy to clean the pleural space and leave a chest tube postoperatively to drainage. The other group will undergo chest tube placement with subsequent infusion of fibrinolytics to dissolve the thick purulent material allowing drainage.

Both groups will have the same antibiotic regimen with the same management algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years of age requiring an intervention for empyema by one of the following:

  1. Septation or loculation seen on ultrasound or computed tomography
  2. Many white blood cells, bacteria present, or thick viscid purulence identified on pleural tap

Exclusion Criteria:

1. Immunodeficiency process
2. Secondary diagnosis or condition that will keep them in the hospital beyond the empyema
3. Existing contraindications to VATS or chest tube.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization after intervention | 1 month

SECONDARY OUTCOMES:
Days where a maximum temperature was equal to or above 38 degrees C, days of tube drainage, doses of analgesia and days of oxygen requirement, hospital days after intervention, hospital charges after intervention and procedure charges | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States